CLINICAL TRIAL: NCT03593824
Title: The Susceptibility of Phenotypic Plasticity During Adversity and Prosperity in Infants With Visual Deprivation
Brief Title: The Visual Plasticity During Adversity and Prosperity in Infants With Congenital Cataracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Ophthalmologist, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CCPMOH2018-China-6
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Cataract
Keywords: Phenotypic plasticity; Adversity; Prosperity
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dense cataract group (Experimental)
  Interventions: Procedure: bilateral cataract removal surgery for dense cataract
- non-dense nuclear cataract group (Experimental)
  Interventions: Procedure: bilateral cataract removal surgery for non-dense nuclear cataract

INTERVENTIONS:
Procedure: bilateral cataract removal surgery for dense cataract — Participants were born with dense bilateral cataracts (extreme adversity) will undergo surgery for bilateral cataract removal at an early age, mostly around 3 months of age.
  Arms: dense cataract group
Procedure: bilateral cataract removal surgery for non-dense nuclear cataract — Participants were born with non-dense and nuclear bilateral cataracts (watered-down adversity) will undergo cataract removal surgery bilaterally in a compromised timing, mostly around one year old.
  Arms: non-dense nuclear cataract group

SUMMARY:
Phenotypic plasticity is the ability of individuals to change their phenotypic status when exposed to environmental variations. However, whether the plastic changes show differential susceptibility in adversity and prosperity is debated and the specific pattern of plasticity remains elusive.

Here the investigators address this question by tracking the phenotypes (functional, structural, physical, and attachment traits) in two groups of infants before and after visual deprivation: one group experienced a short duration of complete deprivation (extreme adversity) and the other group experienced a long durations of partial deprivation (watered-down adversity).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with dense or non-dense nuclear congenital cataract

Exclusion Criteria:

* no metabolic diseases, mental retardation or central nervous diseases
* had no history of inherited diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in visual acuity measured by Teller visual acuity cards | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months after surgery

SECONDARY OUTCOMES:
Change from baseline in refractive status measured by autorefractor and objective retinoscopy | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ellis BJ, Boyce WT, Belsky J, Bakermans-Kranenburg MJ, van Ijzendoorn MH. Differential susceptibility to the environment: an evolutionary--neurodevelopmental theory. Dev Psychopathol. 2011 Feb;23(1):7-28. doi: 10.1017/S0954579410000611. PMID 21262036
- [Background] Pluess M, Belsky J. Vantage sensitivity: individual differences in response to positive experiences. Psychol Bull. 2013 Jul;139(4):901-16. doi: 10.1037/a0030196. Epub 2012 Oct 1. PMID 23025924